CLINICAL TRIAL: NCT01627587
Title: A Two Cohort, Open-label Study to Evaluate the Pharmacokinetics of GSK2847065, the Metabolite of Retosiban (GSK221149) After Single and Repeat Oral Doses, the Pharmacokinetics of GSK221149 Coadministered With a High Fat Meal, and the Pharmacokinetics of GSK221149 Coadministered With an Inhibitor of CYP3A4 (Ketoconazole)
Brief Title: A Two Cohort Study to Look at the Metabolites of GSK221149, the Metabolism of GSK221149 Administered With a High Fat Meal and With Ketoconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 115893
Record Dates: First submitted 2012-06-14; First posted 2012-06-26 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Obstetric Labour, Premature
Keywords: preterm labor
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Ketoconazole; Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketoconazole-Part A (Experimental): Healthy Female volunteers of child bearing potential will receive Treatment A, B and C
  Interventions: Drug: GSK221149 750 mg; Drug: Ketoconazole; Drug: GSK221149 100 mg
- Food-Part B (Experimental): Healthy Female Volunteers of child bearing potential will receive Treament D and E
  Interventions: Drug: GSK221149 750 mg Fasted; Drug: GSK221149 750 mg + Food

INTERVENTIONS:
Drug: GSK221149 750 mg — Treatment A: 750 mg GSK221149 single dose
  Arms: Ketoconazole-Part A
Drug: Ketoconazole — Treatment B: 400 mg of Ketoconazole single dose
  Arms: Ketoconazole-Part A
Drug: GSK221149 100 mg — Treatment C: 100mg of GSK221149 single dose
  Arms: Ketoconazole-Part A
Drug: GSK221149 750 mg Fasted — Treatment D: 750 mg of GSK221149 administered fasted
  Arms: Food-Part B
Drug: GSK221149 750 mg + Food — Treatment E: 750 mg of GSK221149 administered with a high fat meal
  Arms: Food-Part B

SUMMARY:
This is a two part study. Part A of the study will evaluate the metabolites of GSK221149 following single and repeat oral dosing and will also assess the pharmacokinetics of GSK221149 when administered with a potent CYP3A4 inhibitor Ketoconazole. Part B of the study will look at the pharmacokinetics of GSK221149 following a high fat meal.

ELIGIBILITY:
Inclusion Criteria:

* ALT, alkaline phosphatase and bilirubin less than and equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Single [QTc, QTcB or QTcF] less than 450 msec; or QTc less than 480 msec in subjects with Bundle Branch Block.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Female subjects between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Child-bearing potential and is abstinent or agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 48 hours post last dose.
* Body weight greater than 50 kg and BMI within the range 19-29.9 kg/m2 (inclusive).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol/urine cotinine screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummels, exotic citrus fruits, grapefruit hybrids from 7 days prior to the first dose of study medication.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-12-12 (Actual); Primary Completion 2012-02-09 (Actual); Study Completion 2012-02-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve, half life | From Day 1- Day 11 of the study
Area under the curve, half life, when treate with ketconizole | Day 1-11

SECONDARY OUTCOMES:
12 lead ECGs, safety labs, vital signs, heart rate, blood pressure | Day 1- Day 11 of the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115893 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115893?search=study&study_ids=115893#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 115893 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115893 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115893 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115893 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115893 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115893 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115893 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register